CLINICAL TRIAL: NCT03782389
Title: The Role of Periodic Health Examination in Determining Lower Extremity Muscle Injury Risk in Elite Football (Soccer): A Protocol for an Investigation Into Multivariable Prognostic Model Development, Validation and Prognostic Factor Exploration
Brief Title: The Role of Periodic Health Examination in Determining Indirect Muscle Injury Risk in Elite Football (Soccer)
Status: Completed | Type: Observational
Sponsor: Manchester United Football Club (Other)
Collaborators: University of Manchester (Other); Keele University (Other); Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Tom Hughes, Senior Physiotherapist and Clinical Lead, Manchester United Football Club
Other Study IDs: MUFC1
Record Dates: First submitted 2018-12-12; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Muscle Injury; Sprains and Strains
Keywords: Athlete; injury prevention; muscle strain; prediction; prognosis; screening; sport
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite football players aged 16-40 years
  Interventions: Other: Preseason Periodic Health Examination Completion

INTERVENTIONS:
Other: Preseason Periodic Health Examination Completion — all available players completed a mandatory PHE on one of three days during the first week of the season. Typically, the musculoskeletal and performance components of the PHE included: 1) anthropometric measurements; 2) medical history (i.e. previous injury history); 3) musculoskeletal examination tests; 4) functional movement and balance tests; 5) strength and power tests.

SUMMARY:
Preseason periodic health examination (PHE) is used routinely in elite football (soccer) and can be used to inform injury prevention strategies. Indirect muscle injuries (IMI) are a considerable burden to elite teams. This investigation aims to evaluate whether measurements from PHE can be used in a multivariable model to predict IMI risk in elite players, or to establish prognostic factors that are associated with IMIs.

DETAILED DESCRIPTION:
BACKGROUND Indirect muscle injuries (IMIs) are a considerable burden to elite football (soccer) teams and prevention of these injuries offers many benefits. Preseason medical, musculoskeletal and performance screening (termed periodic health examination (PHE)) is used to help determine players at risk of injuries such as IMIs, where identification of PHE-derived prognostic factors (PF) may inform IMI prevention strategies. Furthermore, using several PFs in combination within a multivariable prognostic model may allow individualised IMI risk estimation and specific targeting of prevention strategies, based upon an individual's PF profile. No such models have been developed in elite football and the current IMI prognostic factor evidence is limited. This study aims to: 1) to develop and internally validate a prognostic model for individualised IMI risk prediction during a season in elite footballers, using the extent of the prognostic evidence and clinical reasoning; 2) explore potential PHE-derived PFs associated with IMI outcomes in elite footballers, using available PHE data from a professional team.

METHODS A retrospective review has been completed of PHE and injury data, routinely collected over 5 years (from 1st July 2013 to 19th May 2018) from a population of elite male players at an English Premier League football club. Of 60 candidate PFs, 15 were excluded. Ten factors will be included in model development, identified from a systematic review, missing data assessment, measurement reliability evaluation and clinical reasoning. A full multivariable logistic regression model will be fitted, to ensure adjustment before backward elimination. The performance and internal validation of the model will be assessed. The remaining 35 candidate PFs are eligible for further exploration, using univariable logistic regression to obtain unadjusted risk estimates. Exploratory PFs will be grouped according to type and incorporated into multivariable logistic regression models to determine risk estimates.

DISCUSSION This study will offer insights into clinical usefulness of a model to predict IMI risk in elite football and highlight the practicalities of model development in this setting. Exploration may identify other relevant PFs for future confirmatory studies, model updating, or influence future injury prevention research.

ELIGIBILITY:
Inclusion Criteria:

* had an outfield position (i.e. not a goalkeeper);
* participated in PHE testing for the relevant season.

Exclusion Criteria:

- if players were on trial or not contracted to the club at the time of PHE.

Ages: 16 Years to 40 Years | Sex: Male
Age Groups: Child, Adult
Study Population: The population under study was of male elite football players aged 16-40 years old at an English Premier League club.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2018-05-19 (Actual); Study Completion 2018-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with an indirect muscle injury. | 11 Months (1 football season)
  Indirect muscle injury defined according to Terminology and Classification of Muscle Injuries Consensus Statement

SECONDARY OUTCOMES:
Number of participants with an indirect muscle injury affecting the hamstring muscle group. | 11 Months (1 football season)
  If there is a sufficient number of outcomes, indirect muscle injuries (defined according to the Terminology and Classification of Muscle Injuries Consensus Statement) that affect the hamstring muscle group may be subgrouped and analysed accordingly.
Number of participants with an indirect structural muscle injury. | 11 Months (1 football season)
  If there is a sufficient number of outcomes, indirect muscle injuries will be categorised into structural injuries (defined as type 3 or 4 injury using the Terminology and Classification of Muscle Injuries Consensus Statement) and analysed accordingly.
Number of participants with an indirect functional muscle injury. | 11 Months (1 football season)
  If sufficient there is a sufficient number of outcomes, indirect muscle injuries will be categorised into functional injuries (defined as type 1a to 2b injuries using the Terminology and Classification of Muscle Injuries Consensus Statement) and analysed accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Riley, PhD, Study Director — Centre for Prognosis Research, Keele University. UK; Jamie Sergeant, PhD, Study Director — Arthritis Research UK Centre for Epidemiology, University of Manchester. UK.; Michael Callaghan, PhD, Study Director — Dept of Health Professions, Manchester Metropolitan University. UK

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes T, Riley R, Callaghan MJ, Sergeant JC. Can prognostic factors for indirect muscle injuries in elite football (soccer) players be identified using data from preseason screening? An exploratory analysis using routinely collected periodic health examination records. BMJ Open. 2023 Jan 24;13(1):e052772. doi: 10.1136/bmjopen-2021-052772. PMID 36693686
- [Derived] Hughes T, Riley RD, Callaghan MJ, Sergeant JC. The Value of Preseason Screening for Injury Prediction: The Development and Internal Validation of a Multivariable Prognostic Model to Predict Indirect Muscle Injury Risk in Elite Football (Soccer) Players. Sports Med Open. 2020 May 27;6(1):22. doi: 10.1186/s40798-020-00249-8. PMID 32462372

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03782389/Prot_SAP_000.pdf